CLINICAL TRIAL: NCT05207709
Title: A Phase III, Multicenter, Open-label Study of Ribociclib vs. Palbociclib in Patients With Advanced Hormone Receptor-positive/HER2-negative/HER2-Enriched Breast Cancer - HARMONIA Trial
Brief Title: Ribociclib vs. Palbociclib in Patients With Advanced Breast Cancer Within the HER2-Enriched Intrinsic Subtype
Acronym: HARMONIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry); Alliance Foundation Trials, LLC. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-2101; 2021-002027-38 (EudraCT Number); LEE011A2303R (Other: Novartis); AFT-58 (Other: Alliance Foundation Trials, LLC)
Record Dates: First submitted 2022-01-04; First posted 2022-01-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Breast Cancer
Keywords: PAM50; intrinsic subtype; HER2-Enriched
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole; Fulvestrant; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ribociclib + Endocrine Therapy (Experimental): Ribociclib + Fulvestrant or Letrozole
  Interventions: Drug: Ribociclib + Letrozole OR Fulvestrant
- Palbociclib + Endocrine Therapy (Experimental): Palbociclib + Fulvestrant or Letrozole
  Interventions: Drug: Palbociclib + Letrozole OR Fulvestrant
- Paclitaxel +/- Tislelizumab - Exploratory cohort (Experimental): Additional experimental Cohort that includes patients with Basal-Like intrinsic subtype.
  Interventions: Drug: Paclitaxel +/- Tislelizumab

INTERVENTIONS:
Drug: Ribociclib + Letrozole OR Fulvestrant — Endocrine Therapy will be selected by the investigator. For premenopausal women and men: LHRH agonist once every 4 weeks
  Arms: Ribociclib + Endocrine Therapy
Drug: Palbociclib + Letrozole OR Fulvestrant — Endocrine Therapy will be selected by the investigator. For premenopausal women and men: LHRH agonist once every 4 weeks
  Arms: Palbociclib + Endocrine Therapy
Drug: Paclitaxel +/- Tislelizumab — Patients in this arm could receive as the first line of therapy
  Arms: Paclitaxel +/- Tislelizumab - Exploratory cohort

SUMMARY:
HARMONIA is an international, multicenter, randomized, open-label and phase III study. The primary objective of this study is to demonstrate that the combination of ribociclib with endocrine therapy (letrozole or fulvestrant) is superior to palbociclib with endocrine therapy (letrozole or fulvestrant) in prolonging progression-free survival in patients with advanced HR+/HER2- and HER2-E breast cancer. The study will enroll approximately 456 patients with HER2-E disease from approximately 95 sites worldwide.

In addition, the HARMONIA trial will include an exploratory cohort of patients with HR+/HER2- and Basal-like disease treated with paclitaxel +/- Tislelizumab. This cohort does not have a predefined sample size and the objective is only exploratory, given the suggested lack of efficacy of the combinations of hormone therapy and CDK4/6 inhibitors in this subgroup of patients. Enrolment into the basal-like cohort will stop once the HER2-E disease cohort is fully enrolled.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically documented HR-positive and HER2-negative breast cancer by local testing
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* advanced (loco regionally recurrent not amenable to curative therapy or metastatic) breast cancer.
* Availability of FFPE tumor block for biomarker analysis, obtained during metastatic period.
* HER2-E or Basal-like subtype as per central PAM50 analysis.
* Measurable disease or non-measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end-organ function
* Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.
* Women of childbearing potential must have confirmed negative serum pregnancy test within 7 days prior to randomization.
* Women of CBP must be willing to use highly effective methods of contraception.
* Patient must have a 6-lead or 12-lead ECG with ALL of the following parameters at screening:

  * QTcF interval (QT interval using Fridericia's correction) at screening < 450 msec.
  * Resting heart rate 50-90 beats per minute (determined from the ECG).

Main Exclusion Criteria:

* Prior therapy with any CDK4/6 inhibitors.
* Patient has received prior treatment with chemotherapy for advanced/metastatic breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 62 months after the first patient enrolled
  using RECIST 1.1 criteria, as assessed by local radiologists/investigators

SECONDARY OUTCOMES:
Progression-free survival 2 | From randomization until documented progression to second line of therapy, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 62 months after the first patient enrolled
  defined as the time from randomization to first documented progression on next-line therapy or death, whichever occurs first
Overall Survival | until patient death, assessed up to approximately 62 months after the first patient enrolled
  the proportion of exitus patients
Overall response and clinical benefit | until disease progression or 24 weeks from treatment start.
  defined as percentage of patients with CR, PR per RECIST 1.1 or SD lasting 24 weeks or longer, as defined by RECIST 1.1.
Time to response and duration of response | time from treatment start to response and time from response to disease progression, assessed up to approximately 62 months after the first patient enrolled
  defined per RECIST 1.1
Adverse events (safety) | from randomization/enrollment to end of study assessed up to approximately 62 months after the first patient enrolled
  Occurrence /severity of AEs, laboratory abnormalities, discontinuation rates, dose reductions/interruptions

CONTACTS AND LOCATIONS:
Overall Officials: Aleix Prat, MD, Principal Investigator — Hospital Clínic of Barcelona / SOLTI; Lisa A Carey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Dan G Stover, MD, Principal Investigator — Stefanie Spielman Comprehensive Breast Center; Tomás Pascual, MD, Principal Investigator — Hospital Clínic of Barcelona / SOLTI cancer research group
Locations (71):
- United States (26):
  - Morton Plant Hospital, Clearwater, Florida
  - University of Miami, Coral Gables, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Mount Sinai Florida, Miami, Florida
  - Northwestern, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Sinai of Baltimore, Baltimore, Maryland
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Baptist Memorial Health Care, Oxford, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - NHOH, Londonderry, New Hampshire
  - Nothwell Health, New York, New York
  - Montefiore, The Bronx, New York
  - University of North Carolina Lineberger, Chapel Hill, North Carolina
  - Novant Health Care, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Dayton Clinical Oncology, Kettering, Ohio
  - Legacy Good Samaritan Hospital and Medical Cente, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - The Medical University of South Carolina, Charleston, South Carolina
  - Upstate Carolina Medical Center, Spartanburg, South Carolina
  - Edwards Comprehensive Cancer Center, Huntington, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Unv. Wisconsin, Madison, Wisconsin
- Portugal (5):
  - Hospital Senhora da Oliveira - Guimarães, Creixomil
  - IPO Lisboa, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - Instituto Portugues de Oncologia de Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar Vila Nova de Gaia, Vila Nova de Gaia
- Spain (40):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Institut Català d' Oncologia (ICO Badalona), Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - IOB-Institute of Oncology. Hospital Quironsalud Barcelona, Barcelona, Barcelona
  - Institut Català d'Oncologia (ICO Hospitalet), L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Institut Català d' Oncologia de Girona (ICO Girona), Girona, Girona
  - Hospital Clínico Universitario de A Coruña, A Coruña, La Coruña
  - Hospital Clínico Universitario de Santiago CHUS, Santiago de Compostela, La Coruña
  - Complejo Asistencial Universitario de León, León, León
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Quiron Salud Sagrado Corazon Sevilla, Seville, Sevilla
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza
  - Hospital General Universitario de Alicante, Alicante
  - Vall d´Hebron University Hospital, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Complejo Hospitalario San Pedro de Alcántara, Cáceres
  - Hospital Universitario Virgen de las Nieves, Granada
  - H. Clínico San Cecilio de Granada, Granada
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Sant Joan de Reus, Reus
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen de la Macarena, Seville
  - Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalinsky K, Accordino MK, Chiuzan C, Mundi PS, Sakach E, Sathe C, Ahn H, Trivedi MS, Novik Y, Tiersten A, Raptis G, Baer LN, Oh SY, Zelnak AB, Wisinski KB, Andreopoulou E, Gradishar WJ, Stringer-Reasor E, Reid SA, O'Dea A, O'Regan R, Crew KD, Hershman DL. Randomized Phase II Trial of Endocrine Therapy With or Without Ribociclib After Progression on Cyclin-Dependent Kinase 4/6 Inhibition in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Metastatic Breast Cancer: MAINTAIN Trial. J Clin Oncol. 2023 Aug 20;41(24):4004-4013. doi: 10.1200/JCO.22.02392. Epub 2023 May 19. PMID 37207300
- See also: Related Info — https://www.gruposolti.org/clinicaltrials/harmonia/?lang=en